CLINICAL TRIAL: NCT06010797
Title: Effect of Pre-treatment Photographs on Oral Hygiene Maintenance in Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rehmat Memorial Post Graduate Dental Teaching Hospital (Other)
Responsible Party: Principal Investigator, Eizza Niaz, Principal Investigator, Rehmat Memorial Post Graduate Dental Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RehmatMPGDTH
Record Dates: First submitted 2023-08-20; First posted 2023-08-25 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Oral Hygiene; Photographs
Keywords: Oral hygiene; Photographs; Dental; Orthodontics; Periodontitis; Gingivitis; Index
MeSH Terms: conditions — Periodontitis; Gingivitis; Erythema Multiforme

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: It was a double blinded randomized controlled trial. Patients and the investigator recording indices were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orthodontic patients who are shown pre-treatment photographs (Experimental): Group A included 30 patients who were shown their pre-treatment extra-oral and intra-oral photographs.
  Interventions: Device: Showing Pre-treatment photographs of the patient
- Orthodontic patients who were not shown pre-treatment photographs (No Intervention): Group B included 30 patients who were not shown their pre-treatment extra-oral and intra-oral photographs.

INTERVENTIONS:
Device: Showing Pre-treatment photographs of the patient — Extra-oral and intra-oral dental photographs of patients were taken before starting Orthodontic treatment. Experimental group were shown their photographs while control group were not shown their photographs.
  Arms: Orthodontic patients who are shown pre-treatment photographs

SUMMARY:
Dental photography is an essential component of orthodontic treatment. Photographs enable the clinician to keep record of different stages of treatment. Other uses are for treatment planning, communicating with the patients and other specialists, comparison of pre-treatment and post-treatment changes, for research purpose and also for patient's motivation. Images captured before, during and after treatment provide legal protection when necessary. In the orthodontic discipline, at least three extra-oral and five intra-oral photographs are recommended. Extra-oral photographs should correctly reflect patient's appearance and intra-oral photographs should show complete dentition and occlusion.

Oral hygiene is controlled by the patient during orthodontic treatment which requires proper motivation. Motivational methods are classified as chair-side education, message reminders, behavioral modification and Hawthorne effect. Patients' motivation plays an important role in maintaining favorable oral hygiene. A number of studies have shown the effect of motivational methods on oral hygiene improvement. In one of these studies, 80 patients who needed orthodontic treatment were selected and randomly distributed into two equal groups as control group and study group. The study group patients were included in a Whatsapp where they shared their own photographs (selfies) and received text messages, while the control group patients were not included in any Whatsapp group. Baseline PI scoring was 0.48(0.34) in control group and 0.41(0.32) in study group, After 3 months PI scoring was 1.72(0.33) in control group and 1.68(0.40) in study group. Results showed that sharing of selfies improves oral hygiene compliance in Orthodontic patients.

The purpose of this study was to determine probable effect of pre-treatment photographs on oral hygiene maintenance in orthodontic patients. To our knowledge no such study has been done previously. This would help us in making patients understand the importance of oral hygiene maintenance. The results will also be used by other practitioners.

DETAILED DESCRIPTION:
Randomized Controlled Trial Design:

1. Participants:

   Orthodontic patients.
2. Intervention:

   Patients' own pre-treatment dental photographs.
3. Study group:

   Orthodontic patients who are shown dental photographs.
4. Comparison group:

   Orthodontic patients who are not shown dental photographs.
5. Outcome:

   Good oral hygiene measured by plaque index.
6. Block randomization:

   To decrease selection or accidental bias patients were assigned group A or B using block randomization technique. Blocks were created, size of each block was 4 with 2 'A's and 2 'B's. For 2 groups there were 6 possible blocks. From random number table a random sequence of blocks was generated. Patients were then assigned groups according to blocks.
7. Subjects:

I. Group 1:

Included 30 patients and these patients were shown full extra-oral and intra-oral photographs.

II. Group 2:

Included 30 patients and these patients were not shown any photographs. All subjects received similar oral hygiene instructions. Those in group A were shown their photographs while those in B were not shown any photographs.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders
* Between age 13-25 years

Exclusion Criteria:

* Patients with previous orthodontic treatment
* Handicapped patients
* Patients with any systemic disease
* Generalized periodontal disease
* Congenital malformations

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-07-04 (Actual); Study Completion 2021-07-04 (Actual)

PRIMARY OUTCOMES:
Good oral hygiene measured by plaque index | 3 months
  Plaque scores at T0 and T1 were compared to assess improvement in oral hygiene

CONTACTS AND LOCATIONS:
Locations (1):
- Rehmat Memorial Dental Postgraduate Teaching Hospital, Abbottabad, Khyber Pakhtaunkha, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-08-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT06010797/Prot_SAP_ICF_000.pdf